CLINICAL TRIAL: NCT06167538
Title: Clinical Outcome Following Early Decannulation of Severe Acquired Brain Injury Patients: a Retrospective Cohort Study
Brief Title: Clinical Outcome Following Early Decannulation of Severe Acquired Brain Injury Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Robbert-Jan van Hooff, Clinical Head, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: p-2023-14366
Record Dates: First submitted 2023-11-17; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Tracheostomy Decannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SABI patients with a tracheal tube treated with the new decannulation procedure.: All adult SABI patients ≥ 18 years with a tracheal tube at admission to the Department of Brain Injury from September 2021 to October 2022 and treated with the new decannulation procedure.
  Interventions: Other: Decannulation
- SABI patients in whom decannulation was attempted before implementation of the new procedure.: Patients with SABI and a tracheal tube in whom decannulation was attempted between July 2019 until December 2020 will serve as a historical control group.
  Interventions: Other: Decannulation

INTERVENTIONS:
Other: Decannulation — From the 1st of September 2021, the investigators started to perform decannulation earlier after admission to the Department of Brain Injury. Before attempting to decannulate a patient, several factors were considered and assessed by the patient's treating team: patient's level of consciousness, hemodynamical stability, need for and frequency of salivary aspiration, cough strength and respiration frequency. Patients could not be under treatment for pneumonia and simultaneously have respiratory instability at the time of decannulation.

SUMMARY:
After severe acquired brain injury (SABI: severe traumatic brain injury, stroke, anoxic brain damage), up to 50-70% of patients are tracheostomized. The need to tracheostomize a patient is based on the prolonged inability to breathe and/or protect their airway sufficiently. This is usually done in an Intensive Care Unit (ICU). A tracheostomy is first removed when the patient's clinical conditions allow for it. The removal can be performed in many settings, a neurological rehabilitation unit being one of these.

The overall objective of this study is to evaluate the safety of this earlier decannulation procedure in patients with SABI at our department as well as the effectiveness on functional ability.

ELIGIBILITY:
Inclusion Criteria:

All severe acquired brain injury patients ≥ 18 years with a tracheal tube at admission.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult SABI patients ≥ 18 years with a tracheal tube at admission to the Department of Brain Injury from September 2021 to October 2022 and treated with the new decannulation procedure will be included. Patients with SABI and a tracheal tube in whom decannulation was attempted between July 2019 until December 2020 will serve as a historical control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at three months after hospital discharge | Three months counted from hospital discharge
  Rate of survival
Mortality at twelve months after hospital discharge | Twelve months counted from hospital discharge
  Rate of survival

SECONDARY OUTCOMES:
Rate of antibiotics prescribed to treat pneumonia after decannulation | Counted number of days from decannulation until discharge
  Pneumonia as assessed by treating physician
Rate of re-cannulation of the tracheal tube after initial decannulation | Counted number of days from decannulation until discharge
  Assessment of failed decannulation attempts
Length of hospital stay | Counted number of days from admission to our department until discharge
  LOS counted from admission to our department
Rate of hospital readmission at two and twelve months after discharge | At two and twelve months respectively counted from discharge
  Rate of hospital readmission, and if yes, for what cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Brain Injury, Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided